CLINICAL TRIAL: NCT02966600
Title: Effects of Progressive Resistance Exercise in Akinetic-rigid Parkinson's Disease Patients
Brief Title: Strength Training and Different Subtypes of Parkinson´s Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Luis Santos, PhD, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UOviedo
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive resistance exercise (PRE) (Experimental): Progressive resistance exercise (PRE) in akinetic-rigid Parkinson's disease patients. Intervention included sixteen PRE training sessions for eight weeks: two sessions per week on non-consecutive days, sixty-seventy min each one.
  Interventions: Other: Progressive resistance exercise; Other: Physical Activity
- Physical Activity (No Intervention): The control group followed its usual weekly physical activity routine

INTERVENTIONS:
Other: Progressive resistance exercise — The intervention group participated in sixteen PRE training sessions for eight weeks: two sessions per week on non-consecutive days, sixty-seventy min each one.
  Arms: Progressive resistance exercise (PRE)
Other: Physical Activity — The control group followed its usual weekly physical activity routine
  Arms: Progressive resistance exercise (PRE)

SUMMARY:
The aim of this randomized controlled trial was to assess the impact of progressive resistance exercise (PRE) in PD patients with akinesia and rigidity (AR-subtype). The investigators hypothesized the intervention would have a beneficial effect on the study outcomes.

DETAILED DESCRIPTION:
Twenty-eight patients with PD AR-type of both sexes, were recruited for this trial. Each participant were assigned randomly to either intervention (N=13) or control (N=15) group.

The intervention group participated in sixteen PRE training sessions for eight weeks: two sessions per week on non-consecutive days, sixty-seventy min each one. The control group followed their usual weekly physical activity routine.

All patients underwent antrophometrical and neuromuscular function assessment (CoP measurements -primary outcomes- and the Ten-Meters Walk Test -TMWT- -secondary outcomes-). In addition, they were asked to provide ratings for the Spanish validated versions of the the Freezing of Gait Questionnaire (FOG-Q, 6-item version) -secondary outcomes-, the 39-item Parkinson ́s disease Questionnaire (PDQ39) -secondary outcomes- and the MDS-UPDRS -secondary outcomes-. Additionally, ratings of perceived exertion (RPE) (Borg >6-20 scale) - secondary outcomes-, were recorded at the end of each PRE training session. Tests were carried out at three times: pre-test (before the training program), post-test (eight weeks after pre-tests, at the end of the training period), and four weeks after the post-test (re-test).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PD AR-type and Hoehn and Yahr Scale 1-2, (H&Y)
* Do not express any type of dementia
* Able to stand for two min without assistance;
* Able to walk ten metres without assistance.

Exclusion criteria:

* To suffer a neurological disease other than PD.
* Do not meet some of the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Static posturography through the centre of pressures measurements (CoP). | Eight weeks

SECONDARY OUTCOMES:
Gait. | Eight weeks
Freezing of gait. | Eight weeks
The Movement Disorders Society-Unified Parkinson ́s Disease Rating Scale. (MDS-UPDRS). | Eight weeks
The patient- perceived quality of life. | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luis Santos, PhD, Principal Investigator — University School of Sports Medicine, University of Oviedo, Spain. Performance and Health Group, Department of Physical Education and Sport. Faculty of Sports Sciences and Physical Education, University of A Coruna, Spain.
Locations (1):
- University School of Sports Medicine, University of Oviedo, Spain., Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886